CLINICAL TRIAL: NCT02050906
Title: The Intensive Diet and Exercise Adherence Trial - Pilot (IDEA-P): A Feasibility Study of a Lifestyle Intervention in Men Undergoing Androgen Deprivation Therapy
Brief Title: Intensive Diet and Exercise or Standard of Care in Improving Physical Function and Quality of Life in Patients With Prostate Cancer Undergoing Androgen Deprivation Therapy
Acronym: IDEA-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OSU-12008; NCI-2013-01328 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R03CA162969 (NIH)
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Prostate Cancer; Stage IV Prostate Cancer
Keywords: IDEA-P; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (diet and exercise intervention) (Experimental): EXERCISE COMPONENT: Patients undergo 1 hour of monitored intensive exercise comprising 30 minutes of aerobic exercise and 30 minutes of resistance exercise twice weekly during weeks 1-6, once weekly during weeks 7-8, and independently during weeks 7-12. All patients will complete a comprehensive exercise and quality-of-life assessment at baseline, month 2 and month 3.
  BEHAVIORAL ACTIVITY COUNSELING: Patients undergo behavioral activity counseling in small group sessions over 20 minutes once weekly during months 1-2 and individualized activity counseling via telephone calls over 20 minutes every 2 weeks for 3 months. Counseling will include questionnaire administration.
  BEHAVIORAL DIETARY INTERVENTION: Patients undergo nutritional counseling over 30 minutes once weekly during months 1-2 and then every 2 weeks via telephone calls during month 3.
  Interventions: Behavioral: behavioral dietary intervention; Behavioral: exercise intervention; Other: behavioral activity counseling; Behavioral: telephone based counseling; Procedure: quality-of-life assessment; Other: questionnaire administration
- Arm II (standard of care) (Active Comparator): TELEPHONE BASED COUNSELING: Patients receive standard care and educational literature describing the American Institute of Cancer Research dietary and physical activity guidelines. Patients also receive phone calls over 20 minutes every 2 weeks for 3 months focusing on routine prostate cancer self-management. After 3 months, patients have the option to undergo 2 supervised exercise training and dietary counseling sessions. All patients will complete a comprehensive exercise and quality-of-life assessment at baseline, month 2 and month 3.
  Interventions: Procedure: quality-of-life assessment; Other: questionnaire administration

INTERVENTIONS:
Behavioral: behavioral dietary intervention — Patients undergo nutritional counseling over 30 minutes once weekly during months 1-2 and then every 2 weeks via telephone calls during month 3.
  Arms: Arm I (diet and exercise intervention)
Behavioral: exercise intervention — Patients undergo 1 hour of intensive exercise comprising 30 minutes of aerobic exercise and 30 minutes of resistance exercise twice weekly during weeks 1-6, once weekly during weeks 7-8, and independently during weeks 7-12.
  Arms: Arm I (diet and exercise intervention)
Other: behavioral activity counseling — Undergo behavioral activity and nutritional counseling
  Other Names: counseling and communications studies
  Arms: Arm I (diet and exercise intervention)
Behavioral: telephone based counseling — Undergo behavioral activity and nutritional counseling
  Arms: Arm I (diet and exercise intervention)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies intensive diet and exercise or standard of care in improving physical function and quality of life in patients with prostate cancer undergoing androgen deprivation therapy. Diet and exercise may help improve physical function and quality of life in prostate cancer patients. It is not yet known whether intensive diet and exercise is more effective than standard of care in improving physical function and quality of life in patients with prostate cancer undergoing androgen deprivation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the effects of the intensive lifestyle intervention and standard of care treatments on functional limitations (FL), body composition (BC), and quality of life (QOL) in prostate cancer (PC) patients on androgen deprivation therapy (ADT).

II. To determine the feasibility of delivering an intensive lifestyle exercise and dietary intervention to PC patients undergoing ADT.

III. To identify the intermediate variables that account for the beneficial effect of the lifestyle intervention on functional limitations and QOL.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I:

EXERCISE COMPONENT: Patients undergo 1 hour of intensive exercise comprising 30 minutes of aerobic exercise and 30 minutes of resistance exercise twice weekly during weeks 1-6, once weekly during weeks 7-8, and independently during weeks 7-12.

BEHAVIORAL ACTIVITY COUNSELING: Patients undergo behavioral activity counseling in small group sessions over 20 minutes once weekly during months 1-2 and individualized activity counseling via telephone calls over 20 minutes every 2 weeks for 3 months.

DIETARY COMPONENT: Patients undergo nutritional counseling over 30 minutes once weekly during months 1-2 and then every 2 weeks via telephone calls during month 3.

ARM II: Patients receive standard care and educational literature describing the American Institute of Cancer Research dietary and physical activity guidelines. Patients also receive phone calls over 20 minutes every 2 weeks for 3 months focusing on routine prostate cancer self-management. After 3 months, patients undergo 2 supervised exercise training and dietary counseling sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PC: histologically-defined diagnosis of PC based upon providing pathology reports and staging studies
* Initiating ADT: will be initiating a planned course of at least 3 months of ADT; the ADT is defined as: (a) surgical castration; (b) gonadotropin-releasing hormone (GNRH) antagonist alone; (c) GNRH antagonist with oral androgen receptor blockade, and (d) GNRH antagonist, oral androgen receptor blockade, and 5-alpha reductase inhibitors; we will not include men with only oral antiandrogen therapy such as 5-alpha reductase inhibitors alone or oral antiandrogens alone, as they do not produce castrate levels of testosterone
* Stage: at enrollment, all men have stage IV disease, which is our major presentation to the medical oncology prostate program; two groups are typical; the first involves men who usually present for initial diagnosis with minimally metastatic disease and elevated prostate-specific antigen (PSA) and staging studies with modest nodal enlargement or bone lesions, typically asymptotic; the second group involves men we have been monitoring after local therapy, surgery or radiation, but who have a slow rise in PSA indicating failure of curative therapy; at some point in time asymptomatic metastases are noted on scans, and ADT is offered
* Sedentary lifestyle: fewer than 60 minutes of participation in structured moderate intensity physical activity each week
* Health status: all participants must be free of active cardiovascular disease (CVD), unstable angina, arrhythmia, or severe systemic disease that would make moderate intensity exercise participation unsafe; men with prior CVD that have had successful intervention/treatment that are no longer have active CVD and are medically cleared to safely exercise by their physician will be eligible to participate in the study
* Consents: willing to give an informed consent and sign a Health Insurance Portability and Accountability Act (HIPPA) authorization form
* Physician medical clearance: all men will have medical clearance to participate in the study from a board certified internist, primary care physician, or cardiologist (for men with ongoing cardiovascular disease) prior to inclusion in the study; all participants' treating oncologists will also provide consent for participation prior to inclusion in the study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05-21 (Actual); Primary Completion 2015-07-29 (Actual); Study Completion 2015-07-29 (Actual)

PRIMARY OUTCOMES:
Change in FL as measured by the abbreviated Late-Life Function, Disability Inventory (LL-FDI), and Mobility-Related Self-Efficacy | Baseline to up to 3 months
  Exploratory analyses of the direct and indirect pathways of the intervention effects on change in FL will be conducted using a structural equation modeling longitudinal panel model approach.
Change in functional performance assessed using the 400 meter walk, stair-climb, and lift and carry task | Baseline to up to 3 months
Change in muscular strength, assessed using standardized one-repetition maximum testing protocols for chest press and leg extension exercises | Baseline to up to 3 months
Change in body composition, assessed using the Bod Pod whole-body air displacement plethysmography system and GE Lunar dual-energy X-ray absorptiometry (iDXA) system | Baseline to up to 3 months
Change in body weight, measured using a calibrated and certified balance beam scale | Baseline to up to 3 months
Change in global and disease-specific QOL assessed using the Satisfaction with Life Scale, the Short Form (SF)-36, and the Functional Assessment of Cancer Treatment-Prostate (FACT-P) | Baseline to up to 3 months
  Exploratory analyses of the direct and indirect pathways of the intervention effects on change in QOL will be conducted using a structural equation modeling longitudinal panel model approach.
Change in pain and fatigue, assessed using the short-form McGill Pain Questionnaire and the Brief Fatigue Inventory (BFI) | Baseline to up to 3 months
Change in physical activity assessed using the Community Healthy Activities Model Program For Seniors (CHAMPS), Leisure-Time Exercise Questionnaires, and LIFECORDER Plus Accelerometer | Baseline to up to 3 months
Change in exercise-related self-efficacy, assessed using Exercise Self-Efficacy, Barrier Self-Efficacy, Multi-dimensional, and Self-Regulatory Self-Efficacy scales | Baseline to up to 3 months
Change in dietary behavior using the Fred Hutchinson Food Frequency Questionnaire and three-day diet records | Baseline to up to 3 months
Feasibility of delivering an intensive lifestyle exercise and dietary intervention, assessed using recruitment rates, intervention adherence, adverse events, and retention rates | Up to 3 months
  Descriptive statistics will be calculated prospectively throughout the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Focht, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Focht BC, Lucas AR, Grainger E, Simpson C, Fairman CM, Thomas-Ahner JM, Chaplow ZL, DeScenza VR, Bowman J, Clinton SK. Effects of a Group-Mediated Cognitive Behavioral Lifestyle Intervention on Select Social Cognitive Outcomes in Prostate Cancer Patients Undergoing Androgen Deprivation Therapy. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419893764. doi: 10.1177/1534735419893764. PMID 31838879
- [Derived] Focht BC, Lucas AR, Grainger E, Simpson C, Fairman CM, Thomas-Ahner JM, Buell J, Monk JP, Mortazavi A, Clinton SK. Effects of a Group-Mediated Exercise and Dietary Intervention in the Treatment of Prostate Cancer Patients Undergoing Androgen Deprivation Therapy: Results From the IDEA-P Trial. Ann Behav Med. 2018 Apr 19;52(5):412-428. doi: 10.1093/abm/kax002. PMID 29684136
- [Derived] Focht BC, Lucas AR, Grainger E, Simpson C, Thomas-Ahner JM, Clinton SK. The Individualized Diet and Exercise Adherence Pilot Trial (IDEA-P) in prostate cancer patients undergoing androgen deprivation therapy: study protocol for a randomized controlled trial. Trials. 2014 Sep 9;15:354. doi: 10.1186/1745-6215-15-354. PMID 25199619
- See also: The Jamesline — http://cancer.osu.edu